CLINICAL TRIAL: NCT02457949
Title: The Impact of Alternative Social Assistance Disbursement on Drug-Related Harm: a Randomized Control Trial
Brief Title: The Impact of Alternative Social Assistance Disbursement on Drug-related Harm
Acronym: TASA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analyses produced signal of intervention efficacy for primary outcomes and weaker signal of increased exposure to violence. Therefore, DSMC recommended stopping recruitment in May 2018. Enrolled participants completed intervention by Aug 2018
Sponsor: University of British Columbia (Other)
Collaborators: BC Centre on Substance Use (Other)
Responsible Party: Principal Investigator, Lindsey Richardson, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H14-02401
Record Dates: First submitted 2015-05-13; First posted 2015-05-29 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Drug Use
Keywords: Social Assistance; Drug Use; Drug-Related harm

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment As Usual (TAU) (No Intervention): Receipt of social assistance on government cheque issue days for 6 income assistance cycles (approx 26 weeks).
- Staggered Arm (Experimental): Receipt of social assistance once monthly on a randomly assigned day that does not fall during the week of government cheque issue (Non-synchronized social assistance receipt), for 6 income assistance cycles (approx 26 weeks).
  Interventions: Other: Non-synchronized social assistance receipt
- Staggered and Split Arm (Experimental): Receipt of social assistance twice monthly on equally spaced randomly assigned days that do not fall during the week of government cheque issue (Non-synchronized social assistance receipt, cheque divided into two equal disbursements), for 6 income assistance cycles (approx 26 weeks).
  Interventions: Other: Non-synchronized social assistance receipt; Other: cheque divided into two equal disbursements

INTERVENTIONS:
Other: Non-synchronized social assistance receipt — Social assistance disbursement outside government cheque issue week
  Other Names: Staggered
  Arms: Staggered Arm; Staggered and Split Arm
Other: cheque divided into two equal disbursements — Social assistance disbursement divided into two equal payments
  Other Names: Split
  Arms: Staggered and Split Arm

SUMMARY:
This study evaluates whether altering the timing and frequency of social assistance disbursement reduces drug related-harms that increase on the days surrounding monthly synchronized government social assistance cheque issue.

DETAILED DESCRIPTION:
Coordinated monthly income assistance payments, while seeking to alleviate poverty, can also have negative and unintended impacts, particularly among people who use illicit drugs (PWUD). Observational research has identified escalations in drug-related harm coinciding with monthly assistance payments, such as overdose, treatment interruption, hospital admissions and public disorder. This project varies the timing and frequency of income assistance disbursement, and evaluates whether varying income assistance disbursement reduces drug-related harm coinciding with coordinated income assistance.

Conducted among 273 PWUD, participants will be allocated for 6 income assistance cycles to a control or one of two intervention arms. Participants in the control arm will receive payments according to the existing monthly government schedule. Participants in the intervention arm will receive their income assistance: (1) monthly on a day different from government cheque issue; or (2) semi-monthly on days different from government cheque issue. The intervention will be evaluated using qualitative and quantitative methods for its impact on drug use and related harms.

ELIGIBILITY:
Inclusion Criteria:

* be ≥19 years of age or older
* reside in greater Vancouver, Canada
* report regular use of illicit drugs other than cannabis
* receive monthly provincial income assistance
* are not currently administered (where cheque issue/money is externally managed)
* be eligible and willing to be a client of the local credit union who will administer the intervention
* report intensified drug use around government cheque issue days
* provide written informed consent
* be willing to comply with study procedures

Exclusion Criteria:

* plan to relocate outside Vancouver
* have plans to discontinue income assistance

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Illicit drug use on government cheque issue days | 26 weeks
  Timeline Follow Back (TLFB) assessed increase of drug use defined as an increase in the frequency of drug use of at least 40% or an increase in the number of drugs used during the 3 days beginning with government cheque issue day, compared to non-cheque issue days.

SECONDARY OUTCOMES:
Illicit drug use on non-government cheque issue days | 26 weeks
  Timeline Follow Back (TLFB) assessed increase of drug use defined as an increase in the frequency of drug use of at least 40% or an increase in the number of drugs used during the 3 days beginning with individual cheque issue day (among intervention participants), compared to non-cheque issue days.
Hospital admissions on government cheque issue days | 26 weeks
  Emergency Department, Emergency Department Mental Health and substance use hospitalizations in the three days beginning with government cheque issue day compared to non-cheque issue days.
Overdose | 26 weeks
  Self-reported non-fatal overdose and hospital record verified fatal overdose on the three days beginning with government cheque issue day compared to non-cheque issue days.
Police service utilization | 26 weeks
  Self-reported and police record-verified interactions with police or use of police services on the three days beginning with government cheque issue day compared to non-cheque issue days.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Richardson, DPhil, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Centre on Substance Use, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Richardson L, Laing A, Choi J, Nosova E, Milloy MJ, Marshall BD, Singer J, Wood E, Kerr T. Effect of alternative income assistance schedules on drug use and drug-related harm: a randomised controlled trial. Lancet Public Health. 2021 May;6(5):e324-e334. doi: 10.1016/S2468-2667(21)00023-2. Epub 2021 Apr 12. PMID 33857455
- [Derived] Mendell J, Richardson L. Integrated knowledge translation to strengthen public policy research: a case study from experimental research on income assistance receipt among people who use drugs. BMC Public Health. 2021 Jan 18;21(1):153. doi: 10.1186/s12889-020-10121-9. PMID 33461522
- [Derived] Richardson L, Laing A, Milloy MJ, Maynard R, Nosyk B, Marshall B, Grafstein E, Daly P, Wood E, Montaner J, Kerr T. Protocol of the impact of alternative social assistance disbursement on drug-related harm (TASA) study: a randomized controlled trial to evaluate changes to payment timing and frequency among people who use illicit drugs. BMC Public Health. 2016 Jul 29;16:668. doi: 10.1186/s12889-016-3304-6. PMID 27473400
- See also: British Columbia Centre on Substance Use — http://www.bccsu.ca/cheque-day-study/